CLINICAL TRIAL: NCT05040620
Title: Effectiveness of Olive Oil Local Application in Decreasing the Period of Alignment Phase in Non Extraction Orthodontic Patients. A Randomized Controlled Clinical Trial.
Brief Title: Effectiveness of Olive Oil Local Application in Orthodontic Patients.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Nasef Abdelhameed, Lecturer of Orthodontics, Faculty of Dentistry, Minia University, Egypt, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 455
Record Dates: First submitted 2020-11-15; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Orthodontic Tooth Movement
Keywords: Orthodontic tooth movement, olive oil
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): controlling group who will receive traditional orthodontic treatment.
- Olive Oil (Experimental): experimental group who will receive the local application of Olive Oil five times daily after teeth brushing
  Interventions: Drug: Olive Oil Topical Oil

INTERVENTIONS:
Drug: Olive Oil Topical Oil — the effect of olive oil local application in decreasing orthodontic alighment phase
  Other Names: olive oil
  Arms: Olive Oil

SUMMARY:
The large body of evidence supports the chemotherapeutic potential of substances found in Olive Oil (OO), acting on different sides, such as inflammation, oxidative damage, and even epigenetic modulation. The consumption of OO should be suggested in a healthy diet instead of other types of oils. It looks worthy, to determine the effect of local application of Olive Oil in decreasing the friction between brackets and wires during orthodontic treatment.

DETAILED DESCRIPTION:
During the orthodontic treatment, the friction between the bracket and the arch-wire could prevent the action of forces required for a particular tooth movement. Studies demonstrated that approximately 12 to 60% of the force used to move a tooth is dissipated in the form of friction. Consequently, a delay could occur in the biological response to orthodontic movement. The most important factors that may have an impact on friction are; the composition of the bracket, the arch-wire alloy, the cross-sectional size of the arch-wire, the type of ligation system and the surface roughness of the bracket-archwire assembly.

In addition to the factors related to the orthodontic appliances, saliva is considered to be a biological variable associated with friction, as it acts as a lubricant during sliding mechanics.This fact should be taken into account in laboratory studies that aim to evaluate the performance of the archwire-bracket combinations. However, in the majority of the research studies, the friction test has been conducted without the use of any lubricant, which does not represent the clinical reality where there is saliva introduced during the movement of the arch-wire on the bracket. To remedy this situation, distilled water has been used as a lubricant. Although in this case the test is conducted in the presence of a lubricant, water does not have the lubricating ability of natural human saliva.

It is well known that oil is a well-known lubricant. But how we can use it to decrease friction between brackets and wires? and which type of oil we can use safely in patient mouth? Olive oil (OO) (Olea europaea, Oleaceae) is a fundamental component of the Mediterranean Diet; it is a mix of fatty acids such as oleic and linoleic acid, secoiridoids (oleuropein and oleocanthal), simple phenols (tyrosol and hydroxytyrosol), lignans (pinoresinol), flavonoids (apigenin), hydrocarbons (squalene), triterpenes (maslinic acid), and phytosterols (β-sitosterol).

The large body of evidence supports the chemotherapeutic potential of substances found in OO, acting on different sides, such as inflammation, oxidative damage, and even epigenetic modulation. The consumption of OO should be suggested in a healthy diet instead of other types of oils. It looks worthy, to determine the effect of local application of Olive Oil in decreasing the friction between brackets and wires during orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The age of patients ranges from 15-20 years old.
2. Mild to moderate dental irregularity requiring non-extraction treatment.
3. Presence of all the permanent teeth at least up to the first molars.
4. Good oral hygiene, and periodontal health.

Exclusion Criteria:

1. Patients require orthognathic surgery to correct skeletal discrepancies.
2. patients who are taking medications, like NSAIDs or other anti-inflammatory drugs.
3. cleft lip or palate patients.
4. patients with hypodontia, or hyperdontia.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
The duration of orthodontic teeth aligning using Little irregualrity index | 4 months
  To detect the effect of local usage of Olive Oil on orthodontic brackets during the alignment phase of orthodontic treatment in changing the Little's irregularity in- dex.

SECONDARY OUTCOMES:
orthodontic wire surface roughness changes | one month
  To examine the change in surface roughness of Nickel-Titanium and stainless steel archwires when using Olive Oil as a lubricant and without usage of a lubricant.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nasef, lecturer, Principal Investigator — lecturer of orthodontics, Minia University
Locations (1):
- Ahmed Nasef, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
planning not to share study methodology until finishing the study

REFERENCES:
- [Result] Ehsani S, Mandich MA, El-Bialy TH, Flores-Mir C. Frictional resistance in self-ligating orthodontic brackets and conventionally ligated brackets. A systematic review. Angle Orthod. 2009 May;79(3):592-601. doi: 10.2319/060208-288.1. PMID 19413397
- [Result] Chimenti C, Franchi L, Di Giuseppe MG, Lucci M. Friction of orthodontic elastomeric ligatures with different dimensions. Angle Orthod. 2005 May;75(3):421-5. doi: 10.1043/0003-3219(2005)75[421:FOOELW]2.0.CO;2. PMID 15898384
- [Result] Carrion-Vilches FJ, Bermudez MD, Fructuoso P. Static and kinetic friction force and surface roughness of different archwire-bracket sliding contacts. Dent Mater J. 2015;34(5):648-53. doi: 10.4012/dmj.2014-295. PMID 26438988
- [Result] Matarese G, Nucera R, Militi A, Mazza M, Portelli M, Festa F, Cordasco G. Evaluation of frictional forces during dental alignment: an experimental model with 3 nonleveled brackets. Am J Orthod Dentofacial Orthop. 2008 May;133(5):708-15. doi: 10.1016/j.ajodo.2006.06.021. PMID 18456144
- [Result] Yanase Y, Ioi H, Nishioka M, Takahashi I. Effects of sliding velocity on friction: an in vitro study at extremely low sliding velocity approximating orthodontic tooth movement. Angle Orthod. 2014 May;84(3):451-8. doi: 10.2319/060513-427.1. Epub 2013 Oct 25. PMID 24160997
- [Result] Gorzynik-Debicka M, Przychodzen P, Cappello F, Kuban-Jankowska A, Marino Gammazza A, Knap N, Wozniak M, Gorska-Ponikowska M. Potential Health Benefits of Olive Oil and Plant Polyphenols. Int J Mol Sci. 2018 Feb 28;19(3):686. doi: 10.3390/ijms19030686. PMID 29495598
- [Result] Gotsis E, Anagnostis P, Mariolis A, Vlachou A, Katsiki N, Karagiannis A. Health benefits of the Mediterranean Diet: an update of research over the last 5 years. Angiology. 2015 Apr;66(4):304-18. doi: 10.1177/0003319714532169. Epub 2014 Apr 27. PMID 24778424
- [Result] Curto A, Albaladejo A, Montero J, Alvarado A. Influence of a Lubricating Gel (Orthospeed(R)) on Pain and Oral Health-Related Quality of Life in Orthodontic Patients during Initial Therapy with Conventional and Low-Friction Brackets: A Prospective Randomized Clinical Trial. J Clin Med. 2020 May 14;9(5):1474. doi: 10.3390/jcm9051474. PMID 32423007
- [Result] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05040620/Prot_ICF_000.pdf